CLINICAL TRIAL: NCT04992962
Title: A Double-Blind, Randomized, Placebo-Controlled, Three-Arm Trial Examining Sublingual Cannabinoid Tablets for the Treatment of Pain From Osteoarthritis of the Knee.
Brief Title: Cannabinoid Tablets for the Treatment of Pain From Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pure Green (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG-OA-2021
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
Keywords: CBD; Cannabidiol; CBN; Cannabinol; THC; Osteoarthritis; Pain; Placebo
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD/CBN (Experimental): Participants will receive a 28-day supply of CBD/CBN sublingual tablets to be taken 3 times a day for 28 days.
  Interventions: Drug: CBD/CBN
- CBD/THC (Experimental): Participants will receive a 28-day supply of CBD/THC sublingual tablets to be taken 3 times a day for 28 days.
  Interventions: Drug: CBD/THC
- Placebo (Placebo Comparator): A placebo sublingual tablet to be taken three times a day for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD/CBN — A water-soluble sublingual tablet containing 10 mg of CBD and 10 mg of CBN.
  Arms: CBD/CBN
Drug: CBD/THC — A water-soluble sublingual tablet containing 10 mg of CBD and 5 mg of THC.
  Arms: CBD/THC
Drug: Placebo — An inactive compound.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of PG-OA-10CN and PG-OA-5TH tablets as a better pain reliever in patients with moderate to severe chronic pain due to osteoarthritis of the knee than a placebo.

DETAILED DESCRIPTION:
Subjects will be enrolled in the study for a maximum of 36 days, including a 7-day screening period, 28 days of active product administration, and followed by a post-treatment follow-up within 1 day.

The primary objective of this study is:

* To evaluate the efficacy of PG-OA-10CN and PG-OA-5TH for the treatment of pain associated with osteoarthritis of the knee, compared to a placebo control.

The secondary objectives of this study are:

* To evaluate differences of efficacy between PG-OA-10CN and PG-OA-5TH
* To evaluate the impact of PG-OA-10CN and PG-OA-5TH for stiffness, function in daily living, function in sport and recreation, and knee related quality of life as assessed by the KOOS.
* To evaluate the safety of PG-OA-10CN and PG-OA-5TH for the treatment of pain associated with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 21 years of age;
2. Subject has a diagnosis of osteoarthritis of the knee as determined by the subject's primary care physician or related health care provider.
3. Subject reports an average NPRS score of ≥ 5 in the 7 days prior to enrollment.
4. If female, the subject is postmenopausal (> 1 year), surgically sterile (> 3 months), had a hysterectomy, or is currently using 2 effective forms of birth control.
5. Subject has not taken marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and agrees to not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study.
6. If subject is currently taking a prohibited medication, subject must be willing to and complete a washout of these medications during the screening period and prior to starting study treatment.
7. Subject has not taken any NSAIDs and/or acetaminophen for at least 2 days prior to starting study treatment.
8. Subject is willing to provide his/her written informed consent to participate in the study as stated in the informed consent document.
9. Subject is willing to use an electronic diary to enter trial information for 29 days.

Exclusion Criteria:

1. Subject is pregnant or lactating;
2. Subject has an allergy to cannabis, the Cannabaceae plant family (e.g., hemp, hops), palmitoylethanolamide, or terpenes;
3. Subject has a known allergy to active or inert ingredients of the investigational product;
4. Subject is taking a concomitant medication or treatment that would complicate use or interpretation of the study drug's effects (examples include: Cannabis or any cannabinoid products; Any drug or herbal product that influences the endocannabinoid system (ECS));
5. Subject is taking marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and does not promise that they will not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study;
6. Subject is currently being treated with antibiotics for sinus, throat, or lung infections;
7. Subject has shortness of breath associated with allergies;
8. Subject has uncontrolled asthma;
9. Subject has a fever and/or productive cough;
10. Subject has unstable angina, uncontrolled hypertension;
11. Subject currently or has a history of congestive heart failure;
12. Subject has any other unstable medical condition;
13. Subject has a personal or family history of schizophrenia;
14. Subject has a personal history or currently has suicidal ideation or attempted suicide;
15. Subject has a major neurological disorder, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain injury/head injury, and seizures.
16. Subject has taken pharmaceutical pain medicine, including OTC pain medicine of any kind, or has taken a NSAID and/or acetaminophen within 2 days of starting study treatment.
17. Subject has taken a prohibited medication during the screening period and prior to starting study treatment or is unwilling to stop these medications.
18. Subject has an allergy to, or has an intolerance to, NSAIDs or acetaminophen.
19. Subject has taken any form of steroids, including a local steroid injection in the knee, within 1 month of starting study treatment.
20. Subject has received any invasive interventions or surgery of the knee.
21. Subject has a history of substance or alcohol abuse.
22. Subject has clinically significant illness, including cardiovascular disorders.
23. Subject has any condition in which the investigator believes will confound the data of the study or could put the subject at risk of harm.
24. Subject does not have access to a smart phone or does not know how to use a smart phone application.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-11-14 (Estimated)

PRIMARY OUTCOMES:
Pain as assessed by Numerical Pain Rating Scale (NPRS) | 28 Days
  To evaluate the impact of PG-OA-10CN and PG-OA-10TC on the subject's osteoarthritis of the knee pain as assessed by utilizing a Numeric Pain Rating Scale (NPRS). NPRS is from 0-10, where higher scores indicate worse pain and lower scores indicate less pain reported by the subject.
Pain as assessed by the Knee Injury and Osteoarthritis Outcome Score (KOOS) | 28 Days
  To evaluate the impact of PG-OA-10CN and PG-OA-10TC on the subject's osteoarthritis of the knee pain as assessed by the Knee Injury and Osteoarthritis Outcome Score (KOOS). KOOS is scored from 0-100, where 0 represents extreme problems and 100 represents no problems, as reported by the subject.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events as assessed by CTCAE v4.0. | 28 Days
  To evaluate the safety of PG-OA-10CN and PG-OA-10TC for the treatment of pain associated with osteoarthritis of the knee compared to a placebo control assessed by Common Terminology Criteria For Adverse Events (CTCAE) v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kimless, M.D., Principal Investigator — Pure Green Pharmaceuticals
Locations (1):
- Pure Green Pharmaceuticals, West Bloomfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papaleontiou M, Henderson CR Jr, Turner BJ, Moore AA, Olkhovskaya Y, Amanfo L, Reid MC. Outcomes associated with opioid use in the treatment of chronic noncancer pain in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2010 Jul;58(7):1353-69. doi: 10.1111/j.1532-5415.2010.02920.x. Epub 2010 Jun 1. PMID 20533971
- [Background] Eli Lilly & Company. (2019). Cymbalta: Highlights of prescribing information. Indianapolis, IN.
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Ahrnsbrak, R., Bose, J., Hedden, S. L., Lipari, R. N., & Park-Lee, E. (2017). Key substance use and mental health indicators in the United States: Results from the 2016 National Survey on Drug Use and Health. Center for Behavioral Health Statistics and Quality, Substance Abuse and Mental Health Services Administration, 1572.
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Frakes EP, Risser RC, Ball TD, Hochberg MC, Wohlreich MM. Duloxetine added to oral nonsteroidal anti-inflammatory drugs for treatment of knee pain due to osteoarthritis: results of a randomized, double-blind, placebo-controlled trial. Curr Med Res Opin. 2011 Dec;27(12):2361-72. doi: 10.1185/03007995.2011.633502. Epub 2011 Nov 9. PMID 22017192
- [Background] Blake DR, Robson P, Ho M, Jubb RW, McCabe CS. Preliminary assessment of the efficacy, tolerability and safety of a cannabis-based medicine (Sativex) in the treatment of pain caused by rheumatoid arthritis. Rheumatology (Oxford). 2006 Jan;45(1):50-2. doi: 10.1093/rheumatology/kei183. Epub 2005 Nov 9. PMID 16282192
- [Background] Wang T, Collet JP, Shapiro S, Ware MA. Adverse effects of medical cannabinoids: a systematic review. CMAJ. 2008 Jun 17;178(13):1669-78. doi: 10.1503/cmaj.071178. PMID 18559804
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Michener LA, Snyder AR, Leggin BG. Responsiveness of the numeric pain rating scale in patients with shoulder pain and the effect of surgical status. J Sport Rehabil. 2011 Feb;20(1):115-28. doi: 10.1123/jsr.20.1.115. PMID 21411827
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Ogura T, Ackermann J, Mestriner AB, Merkely G, Gomoll AH. The Minimal Clinically Important Difference and Substantial Clinical Benefit in the Patient-Reported Outcome Measures of Patients Undergoing Osteochondral Allograft Transplantation in the Knee. Cartilage. 2021 Jan;12(1):42-50. doi: 10.1177/1947603518812552. Epub 2018 Nov 22. PMID 30463426
- [Background] Jacquet C, Pioger C, Khakha R, Steltzlen C, Kley K, Pujol N, Ollivier M. Evaluation of the "Minimal Clinically Important Difference" (MCID) of the KOOS, KSS and SF-12 scores after open-wedge high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2021 Mar;29(3):820-826. doi: 10.1007/s00167-020-06026-0. Epub 2020 Apr 27. PMID 32342141